CLINICAL TRIAL: NCT00572572
Title: Phase III, Double-Blind, Placebo-Controlled, Crossover Study Evaluating Aprepitant in Combination With a 5HT3 & Dexamethasone in Patients With Germ Cell Tumors Undergoing 5 Day Cisplatin-Based Chemotherapy Regimen
Brief Title: Aprepitant + a 5HT3 + Dexamethasone in Patients With Germ Cell Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: QL05-37
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Germ Cell Tumors
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Aprepitant, Then Placebo (Experimental): Participants first received Aprepitant 125mg PO day 3 then 80mg on days 4 and 7 during study cycle 1, then received matched placebo PO daily on days 3 through 7 during study cycle 2
  Interventions: Drug: Aprepitant; Drug: Placebo
- Arm B: Placebo, Then Aprepitant (Experimental): Participants first received matched placebo PO daily on days 3 through 7 during study cycle 1, then received Aprepitant 125mg PO day 3 then 80mg on days 4 and 7 during study cycle 2
  Interventions: Drug: Aprepitant; Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — Subjects will be randomized to receive aprepitant 125mg PO day 3 then 80mg on days 4-7 on either cycle 1 or cycle 2.
Drug: Placebo — Subjects will be randomized to receive placebo on days 3-7 on either cycle 1 or cycle 2.

SUMMARY:
Aprepitant is currently approved for prophylaxis of acute and delayed CINV for highly emetogenic chemotherapy regimens, including cisplatin; however, it has not yet been studied in multiple-day chemotherapy treatment programs. This study will compare the addition of aprepitant compared to placebo administered on days 3,4,5 of chemotherapy administration for acute CINV prophylaxis with standard antiemetic prophylaxis and days 6 and 7 for delayed CINV prophylaxis in a double-blind, randomized, crossover study design.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center trial.

Subjects will be stratified prior to randomization based on previous administration of chemotherapy.

Subjects will randomize to aprepitant or placebo with their first study cycle of chemotherapy and then cross over to opposite treatment with the second study cycle.

Cisplatin-based regimen for germ cell tumors containing 20mg/m2/day IV days 1 through 5, first day of chemotherapy administration is day 1. Permitted treatment regimens:

Regimen 1 (BEP) Cisplatin (20mg/m2/day) IV on days 1 to 5 Etoposide (100 mg/m2/day) IV on days 1 to 5 Bleomycin 30 U/IV on days 1, 8, 15

Regimen 2 (EP) Cisplatin (20mg/m2/day) IV on days 1 to 5 Etoposide (100 mg/m2/day) IV on days 1 to 5

Regimen 3 (VIP) Cisplatin (20mg/m2/day) IV on days 1 to 5 Ifosfamide (1200 mg/m2/day) IV on days 1 to 5 (with mesna uroprophylaxis at 100% ifosfamide dosing) Etoposide (75 mg/m2/day) IV on days 1 to 5

Regimen 4 (VeIP) Cisplatin (20mg/m2/day) IV on days 1 to 5 Ifosfamide (1200 mg/m2/day) IV on days 1 to 5 (with mesna uroprophylaxis at 100% ifosfamide dosing) Vinblastine (0.11 mg/kg/day) IV on days 1 and 2

Regimen 5 (EC) Cisplatin (20mg/m2/day) IV on days 1 to 5 Epirubicin (90 mg/m2/day) IV on day 1

Patients are treated on study for two cycles. At the completion of protocol therapy patients will receive additional chemotherapy at the discretion of the treating investigator.

If a patient requires discontinuation of one medication or more on a regimen, the patient must be discontinued from the study.

Performance Status:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin < 3 x upper limit of normal
* Aspartate aminotransferase (AST, SGOT) < 3 x upper limit of normal
* Alanine aminotransferase (ALT, SGPT) < 3 x upper limit of normal
* Alk Phos < 3 x upper limit of normal

Renal:

* Serum Creatinine <2 mg/dL

Pulmonary:

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histologic, serologic or clinical evidence of germ cell tumor.
* Patients scheduled to receive a 5 day fractionated cisplatin-based combination chemotherapy on permitted regimens
* Prior chemotherapy is allowed. Patients will be stratified based on previous treatment.
* Male patients 15 years of age or older at time of registration.
* Patient will provide written informed consent and authorization to release personal health information.

Exclusion Criteria:

* No known history of anticipatory nausea or vomiting.
* No use of another antiemetic agent within 72 hours prior to beginning chemotherapy.
* No known central nervous system (CNS) metastasis.
* No known hypersensitivity to any component of study regimen.
* No concurrent participation in a clinical trial which involves another investigational agent.
* No use of warfarin while on study.
* No use of agents expected to induce the metabolism of aprepitant which include: Rifampin, Rifabutin, Phenytoin, Carbamazepine, and barbiturates.
* No use of agents which may impair metabolism of aprepitant which include: Cisapride, macrolide antibiotics (Erythromycin, Clarithromycin, Azithromycin), azole antifungal agents (Ketoconazole, Itraconazole, Voriconazole, Fluconazole), Amifostine, Nelfinavir and Ritonavir.

Min Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Einhorn, M.D., Study Chair — Hoosier Oncology Group, Inc.
Locations (6):
- United States (6):
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Siteman Cancer Center, St Louis, Missouri
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Froedtert/Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Albany C, Brames MJ, Fausel C, Johnson CS, Picus J, Einhorn LH. Randomized, double-blind, placebo-controlled, phase III cross-over study evaluating the oral neurokinin-1 antagonist aprepitant in combination with a 5HT3 receptor antagonist and dexamethasone in patients with germ cell tumors receiving 5-day cisplatin combination chemotherapy regimens: a hoosier oncology group study. J Clin Oncol. 2012 Nov 10;30(32):3998-4003. doi: 10.1200/JCO.2011.39.5558. Epub 2012 Aug 20. PMID 22915652
- See also: Hoosier Oncology Group Home Page — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Aprepitant, Then Placebo | Arm B: Placebo, Then Aprepitant
Started | 35 | 34
Completed | 32 | 28
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Aprepitant, Then Placebo | Arm B: Placebo, Then Aprepitant | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Median (Standard Deviation); unit: years] — Median age was specifically reported by the investigator.
  years | 34 (11.2) | 30 (8.6) | 31 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 35 | 34 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 34 | 33 | 67
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 35 | 32 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69
Prior Therapies [Number; unit: participants]
  No Prior Therapy | 29 | 28 | 57
  Chemotherapy Multiple Agent Systemic (CMAS) | 5 | 5 | 10
  CMAS and Surgery | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response.
Description: Participants were followed for chemotherapy induced nausea and vomiting (CINV) through day 8 of cycle 2. Complete response is defined as no emetic episodes and no use of rescue medication.
Time Frame: Participants were evaluated from start of treatment through day 8 of cycle 2.
Measure: Number; unit: percentage of evaluable subjects
Groups:
- Aprepitant: Aprepitant cycle whether aprepitant then placebo or placebo then aprepitant
- Placebo: Placebo cycle whether placebo then aprepitant or aprepitant then placebo
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 60 | 60
percentage of evaluable subjects | 47 | 15

2. Secondary Outcome: Proportion of Patients With no Emesis During the Acute CINV Time Period (Cycle Days 1-5)
Description: Proportion of patients with no emesis regardless of use of rescue medication during cycle days 1-5.
Time Frame: Participants were evaluated from cycle days 1-5.
Measure: Number; unit: percentage of evaluable subjects
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 60 | 60
percentage of evaluable subjects | 80 | 52

3. Secondary Outcome: Proportion of Patients With no Emesis During the Delayed CINV Time Period (Cycle Days 6-8)
Description: Proportion of patients with no emesis regardless of use of rescue medication during cycle days 6-8.
Time Frame: Participants were evaluated from cycle days 6-8.
Measure: Number; unit: percentage of evaluable subjects
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 60 | 60
percentage of evaluable subjects | 92 | 78

4. Secondary Outcome: Visual Analouge (VAS) 100mm Scale Score
Description: The Visual Analouge (VAS) 100mm Scale Score for Chemotherapy Induced Nausea and Vomiting (CINV). Participants were asked to mark a linear scale 100mm in length representing their level of nausea with 0mm indicating no nausea and 100mm indicating severe nausea. The mean VAS scores for days 1-8 combined, by treatment (Aprepitant vs. Placebo) were reported.
Time Frame: Days 1-8
Population: There were 54 subjects during the Aprepitant treatment and 61 subjects during the Placebo treatment for days 1-8 that had complete data for the analysis of the visual analouge scale for nausea and vomiting.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 54 | 61
mm | 22.6 (18.7) | 27.1 (22.1)

5. Secondary Outcome: MD Anderson Symptom Inventory Score
Description: The MD Anderson Symptom Inventory (MDASI) is a brief measure of the severity and impact of cancer-related symptoms. Thirteen core items measure the severity of symptoms and six additional items measure the impact of symptoms. All items are rated on a scale from 0 (not present or did not interfere) to 10 (maximal severity or interference). The mean value of the total nineteen items ranges from 0 to 10.
Time Frame: Days 1-8
Population: There were 64 subjects during the Aprepitant treatment and 62 subjects during the Placebo treatment for days 1-8 that had complete data for the analysis of the M.D. Anderson Symptom Inventory. The mean MDASI scores for days 1-8 combined, by treatment (Aprepitant vs. Placebo) were reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 64 | 62
units on a scale | 3.2 (3.4) | 2.9 (2.6)

6. Secondary Outcome: Preferred Treatment Cycle
Description: Participants were asked which treatment cycles was preferable - aprepitant or placebo cycle.
Time Frame: 2 months
Population: There were 49 subjects during the Aprepitant treatment and the Placebo treatment for each cycle that had complete data for the analysis of the preferred treatment cycle.
Measure: Number; unit: percentage of subjects with a preference
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 49 | 49
percentage of subjects with a preference | 78 | 22

ADVERSE EVENTS:
Groups:
- Aprepitant, Then Placebo: Arm A, Study Cycle 1
  Arm B, Study Cycle 2
  Aprepitant: Aprepitant 125mg PO day 3 then 80mg on days 4 through 7
  Subjects will be stratified prior to randomization based on previous administration of chemotherapy.
  Subjects will randomize to aprepitant versus placebo with their first study cycle of chemotherapy and then cross over to opposite arm with the second study cycle.
  Arm A, Study Cycle 1
  Arm B, Study Cycle 2
- Placebo, Then Aprepitant.: Arm A, Study Cycle 2
  Arm B, Study Cycle 1
  Placebo: Matched placebo PO daily on days 3 through 7
  Subjects will be stratified prior to randomization based on previous administration of chemotherapy.
  Subjects will randomize to aprepitant versus placebo with their first study cycle of chemotherapy and then cross over to opposite arm with the second study cycle.
  Arm A, Study Cycle 2
  Arm B, Study Cycle 1
Arm/Group | Aprepitant, Then Placebo | Placebo, Then Aprepitant.
Serious Adverse Events (participants affected / at risk) | 7/35 | 9/34
Other Adverse Events (participants affected / at risk) | 34/35 | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant, Then Placebo (N=35) | Placebo, Then Aprepitant. (N=34)
CARDIAC ISCHEMIA/INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
COLITIS, INFECTIOUS (E.G., CLOSTRIDIUM DIFFICILE) (Gastrointestinal disorders) | 0 (0) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA(ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 1 (1) | 1 (1)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (1) | 0 (0)
INFECTION (ANC <1.0 X 10E9/L) / VEIN (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 0 (0) | 1 (1)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
THROMBOSIS/EMBOLISM (VASCULAR ACCESS-RELATED) (Vascular disorders) | 1 (1) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant, Then Placebo (N=35) | Placebo, Then Aprepitant. (N=34)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 1 (1) | 2 (2)
ALKALINE PHOSPHATASE (Investigations) | 3 (3) | 2 (2)
ALLERGY/IMMUNOLOGY - OTHER (SPECIFY, __) (Immune system disorders) | 2 (2) | 0 (0)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 5 (6) | 3 (4)
ANOREXIA (Gastrointestinal disorders) | 9 (12) | 8 (8)
APNEA (Psychiatric disorders) | 1 (1) | 0 (0)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 2 (3) | 2 (2)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 1 (1) | 2 (2)
BLOOD/BONE MARROW - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 0 (0) | 1 (4)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 3 (3) | 1 (2)
CARDIAC ARRHYTHMIA - OTHER (SPECIFY, __) (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC GENERAL - OTHER (SPECIFY, __) (Cardiac disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 6 (6) | 13 (14)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
CREATININE (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Gastrointestinal disorders) | 2 (2) | 4 (4)
DENTAL: TEETH (Gastrointestinal disorders) | 0 (0) | 1 (1)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 4 (4) | 5 (6)
DIZZINESS (Nervous system disorders) | 1 (1) | 3 (3)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
EDEMA: HEAD AND NECK (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
EDEMA: LIMB (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 19 (25) | 21 (28)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 4 (4) | 7 (9)
FLUSHING (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 2 (3) | 3 (3)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 3 (4) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 12 (15) | 15 (17)
HEARING: PATIENTS WITHOUT BASELINE AUDIOGRAM AND NOT ENROLLED IN A MONITORING PROGRAM (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 13 (16) | 12 (14)
HEMOGLOBIN (Blood and lymphatic system disorders) | 13 (18) | 7 (9)
HEMORRHAGE, GI / RECTUM (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
HYPERTENSION (Cardiac disorders) | 2 (2) | 0 (0)
ILEUS, GI (FUNCTIONAL OBSTRUCTION OF BOWEL, I.E., NEUROCONSTIPATION) (Gastrointestinal disorders) | 0 (0) | 1 (1)
INFECTION (ANC <1.0 X 10E9/L) / JOINT (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (ANC <1.0 X 10E9/L) / PELVIS NOS (Infections and infestations) | 0 (0) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 1 (1) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LARYNX (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LYMPHATIC (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 1 (1) | 3 (3)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SOFT TISSUE NOS (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / UPPER AIRWAY NOS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / WOUND (Infections and infestations) | 0 (0) | 1 (1)
INSOMNIA (General disorders) | 11 (11) | 12 (14)
JOINT-FUNCTION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 8 (8) | 7 (18)
LIPASE (Investigations) | 1 (1) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 2 (2) | 0 (0)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 9 (10) | 7 (7)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 3 (3) | 3 (3)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 3 (3) | 1 (1)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / STOMACH (Gastrointestinal disorders) | 1 (1) | 0 (0)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 21 (32) | 23 (29)
NEUROLOGY - OTHER (SPECIFY, __) (Nervous system disorders) | 2 (2) | 0 (0)
NEUROPATHY: MOTOR (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY: SENSORY (Nervous system disorders) | 4 (4) | 7 (7)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 12 (20) | 8 (17)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 3 (3) | 2 (2)
PAIN / BACK (General disorders) | 4 (4) | 6 (6)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PAIN / DENTAL/TEETH/PERIDONTAL (Gastrointestinal disorders) | 0 (0) | 2 (2)
PAIN / ESOPHAGUS (Gastrointestinal disorders) | 1 (1) | 1 (1)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
PAIN / HEAD/HEADACHE (General disorders) | 3 (3) | 3 (6)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
PAIN / NECK (General disorders) | 1 (1) | 1 (1)
PAIN / NEURALGIA/PERIPHERAL NERVE (Nervous system disorders) | 0 (0) | 1 (1)
PAIN / PAIN NOS (General disorders) | 1 (1) | 1 (1)
PAIN / PROSTATE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PAIN / RECTUM (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN / SCROTUM (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PAIN / TESTICLE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PAIN / THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
PAIN - OTHER (SPECIFY, __) (General disorders) | 2 (2) | 4 (4)
PHLEBITIS (INCLUDING SUPERFICIAL THROMBOSIS) (Vascular disorders) | 0 (0) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 5 (5) | 8 (15)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Investigations) | 0 (0) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 2 (2) | 0 (0)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RENAL/GENITOURINARY - OTHER (SPECIFY, __) (Renal and urinary disorders) | 1 (1) | 0 (0)
RIGORS/CHILLS (General disorders) | 2 (3) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 1 (1) | 2 (2)
SOMNOLENCE/DEPRESSED LEVEL OF CONSCIOUSNESS (Psychiatric disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
SWEATING (DIAPHORESIS) (General disorders) | 2 (2) | 0 (0)
SYNCOPE (FAINTING) (Nervous system disorders) | 1 (1) | 0 (0)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 5 (7) | 2 (2)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 6 (6) | 3 (3)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
TRIGLYCERIDE, SERUM-HIGH (HYPERTRIGLYCERIDEMIA) (Investigations) | 1 (1) | 0 (0)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 8 (9) | 14 (19)
WEIGHT GAIN (General disorders) | 3 (3) | 3 (3)
WEIGHT LOSS (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No